CLINICAL TRIAL: NCT00266812
Title: Randomized Phase II Study: Temozolomide (TMZ) Concomitant to Radiotherapy Followed by Sequential TMZ in Advanced Non-Small Cell Lung Cancer (NSCLC) Patients With Central Nervous System (CNS) Metastasis Versus Radiotherapy Alone
Brief Title: Safety and Tolerability of Low-Dose Temozolomide During Whole Brain Radiation in Patients With Cerebral Metastases From Non-Small-Cell Lung Cancer (Study P04071)(TERMINATED)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Patient target could not be reached within the planned timeframe.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: AESCA Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04071
Record Dates: First submitted 2005-12-16; First posted 2005-12-19 (Estimated); Results first posted 2009-09-04 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: temozolomide; radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemotherapy with temozolomide and radiotherapy (Experimental)
  Interventions: Drug: Temozolomide and radiotherapy
- Radiotherapy alone (Active Comparator)
  Interventions: Procedure: Whole brain radiotherapy

INTERVENTIONS:
Drug: Temozolomide and radiotherapy — Oral temozolomide 75mg/m2/day for 14 days, during radiation treatment, and later on temozolomide 100 mg/m2/day at 14 days on/14 days off, until unacceptable toxicity or evidence of disease progression for up to 6 cycles from initial treatment. Radiotherapy (as in Intervention 2).
  Other Names: Temodal, TMZ, SCH 052365
  Arms: Chemotherapy with temozolomide and radiotherapy
Procedure: Whole brain radiotherapy — 2 regimens are allowed: a) 20 fractions of 2 Gray each, administered on days 1 to 5, 8 to 12, 15 to 19, and 22 to 26; b) 10 fractions of 3 Gray each, administered on days 1 to 5 and 8 to 12.
  Arms: Radiotherapy alone

SUMMARY:
This is a phase II, randomized, multicenter, open-label study designed to assess the safety and tolerability of concomitant chemotherapy with low-dose temozolomide during whole brain radiation and later on at 14 days on/14 days off schedule in patients with cerebral metastases from non-small cell lung cancer (NSCLC). The response to temozolomide will be evaluated by clinical follow up and Magnetic Resonance Imaging (MRI) performed every 2 months. Progression-free survival at 6 months, duration of overall survival, and quality of life will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Prior histologic confirmation of non-small cell lung cancer (NSCLC).
* Optional: NSCLC histologic confirmation of metastasis of NSCLC.
* Presence of unidimensionally measurable disease in the brain.
* No previous or current malignancies at other sites with the exception of adequately treated in situ carcinoma of the cervix or basal and squamous carcinoma of the skin.
* Age: >18 years.
* Subjects must not have systemic disease that in the opinion of the investigator is in immediate need of chemotherapy
* Karnofsky Performance status >=70%.
* Absolute neutrophil count (ANC) >1,500/mm^3, platelets >100,000/mm^3, hemoglobin >8 g/dL.
* Serum creatinine and bilirubin <1.5 times upper normal limit of testing laboratory.
* Serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT) <3 times upper limit of testing laboratory.
* Palliative radiation therapy to thorax and bone or other organs (except brain) is acceptable.
* Prior neurosurgery >2 weeks from initiating treatment with temozolomide.
* Cortisone medication stable or decreasing within 2 weeks prior to initiating treatment with temozolomide.
* Patient is not pregnant or nursing and is advised and willing to use an effective method of contraception.
* Written informed consent.

Exclusion Criteria:

* Chemotherapy or biologic therapy within four weeks prior to initiating therapy with temozolomide.
* Prior radiation therapy for brain <4 weeks from initiating therapy with temozolomide.
* Surgery within two weeks prior to temozolomide administration.
* Recursive Partitioning Analysis (RPA) class III
* Patients with a single brain metastasis amenable to radiosurgery of resection
* Known Human Immunodeficiency Virus (HIV) disease.
* Acute infection requiring intravenous antibiotics.
* Any reason making compliance to the protocol improbable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-03-08 (Actual); Primary Completion 2008-01-16 (Actual); Study Completion 2008-01-16 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy With Temozolomide and Radiotherapy: Oral temozolomide 75mg/m2/day for 14 days, during radiation treatment, and later on temozolomide 100mg/m2/day at 14 days on/14 days off, until unacceptable toxicity or evidence of disease progression for up to 6 cycles from initial treatment. Radiotherapy (as in Intervention 2).
- Radiotherapy Alone: 2 regimens are allowed: a) 20 fractions of 2 Gray each, on days 1 to 5, 8 to 12, 15 to 19, and 22 to 26; b) 10 fractions of 3 Gray each, administered on days 1 to 5 and 8 to 12.
Period: Overall Study
Arm/Group | Chemotherapy With Temozolomide and Radiotherapy | Radiotherapy Alone
Started | 22 | 13
Completed | 1 | 2
Not Completed | 21 | 11
Not completed — Disease Progression | 9 | 3
Not completed — Death | 5 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Discontinued before starting study drug | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy With Temozolomide and Radiotherapy | Radiotherapy Alone | Total
Number analyzed (Participants) | 22 | 13 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.12 (12.72) | 63.02 (8.76) | 64.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 13 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-free Survival (6 Month)
Description: The occurrence of progression will be compared between the study groups by Kaplan-Meier curves. Responsiveness to temozolomide will be evaluated by brain Magnetic Resonance Imanging (MRI)/Computed Tomography (CT), thorax CT, and Quality of Life (QoL) assessments. Progression-free is defined as <25% increase in tumor size on CT or MRI.
Time Frame: 6 months
Population: Intent to treat (ITT) population (31 of the 35 patients enrolled; 4 participants discontinued prior to start of treatment) was analyzed.
Measure: Number; unit: Participants
Arm/Group | Chemotherapy With Temozolomide and Radiotherapy | Radiotherapy Alone
Number analyzed (Participants) | 18 | 13
Participants | 8 | 8

ADVERSE EVENTS:
Arm/Group | Chemotherapy With Temozolomide and Radiotherapy | Radiotherapy Alone
Serious Adverse Events (participants affected / at risk) | 8/18 | 4/13
Other Adverse Events (participants affected / at risk) | 15/18 | 8/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy With Temozolomide and Radiotherapy (N=18) | Radiotherapy Alone (N=13)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 0 (0)
DEATH (General disorders) | 2 (2) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NEOPLASM RECURRENCE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HYDROPNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HOSPITALISATION (Surgical and medical procedures) | 1 (1) | 1 (1)
THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy With Temozolomide and Radiotherapy (N=18) | Radiotherapy Alone (N=13)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 3 (3) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 1 (2) | 0 (0)
DEATH (General disorders) | 1 (1) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 (2) | 0 (0)
PAIN (General disorders) | 1 (1) | 0 (0)
FEBRILE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0)
PYODERMA (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
AGEUSIA (Nervous system disorders) | 1 (1) | 0 (0)
COORDINATION ABNORMAL (Nervous system disorders) | 1 (1) | 0 (0)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 (2) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 1 (1) | 0 (0)
MOTOR DYSFUNCTION (Nervous system disorders) | 2 (2) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (2) | 0 (0)
DEPRESSED MOOD (Psychiatric disorders) | 4 (4) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 2 (2)
DYSSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1)
PERSONALITY CHANGE (Psychiatric disorders) | 1 (1) | 0 (0)
SLEEP DISORDER (Psychiatric disorders) | 2 (2) | 1 (1)
INCONTINENCE (Renal and urinary disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
ECZEMA ASTEATOTIC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
CIRCULATORY COLLAPSE (Vascular disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other